CLINICAL TRIAL: NCT03189160
Title: A Phase 2 Study of Pegylated Recombinant Human Growth Hormone Injection to Treat Children of Turner Syndrome
Brief Title: A Study of PEG-somatropin Injection to Treat Children of Turner Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Beijing Children's Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shanghai Children's Hospital (Other); Children's Hospital of Fudan University (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); The First Hospital of Jilin University (Other); Jiangxi Province Children's Hospital (Other); Affiliated Hospital of Jiangnan University (Other); The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci 032 CT
Record Dates: First submitted 2017-06-13; First posted 2017-06-16 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-06

CONDITIONS: Turner Syndrome
MeSH Terms: conditions — Turner Syndrome | interventions — polyethylene glycol-recombinant human growth hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (3):
- PEG-rhGH low dose (Experimental): PEG-rhGH Injection (27IU/4.5mg/0.5ml/bottle) 0.1 mg/kg/w by subcutaneous injection for 52 weeks.
  Interventions: Biological: PEG-rhGH low dose; Biological: PEG-rhGH high dose; Other: Non-treatment control group
- PEG-rhGH high dose (Experimental): PEG-rhGH Injection (27IU/4.5mg/0.5ml/bottle) 0.2 mg/kg/w by subcutaneous injection for 52 weeks.
  Interventions: Biological: PEG-rhGH low dose; Biological: PEG-rhGH high dose; Other: Non-treatment control group
- Non-treatment control group (No Intervention)

INTERVENTIONS:
Biological: PEG-rhGH low dose — PEG-rhGH Injection 0.1 mg/kg/w by subcutaneous injection for 52 weeks.
  Other Names: Polyethylene Glycol Recombinant Human Somatropin Injection
  Arms: PEG-rhGH high dose; PEG-rhGH low dose
Biological: PEG-rhGH high dose — PEG-rhGH Injection 0.2 mg/kg/w by subcutaneous injection for 52 weeks.
  Other Names: Polyethylene Glycol Recombinant Human Somatropin Injection
  Arms: PEG-rhGH high dose; PEG-rhGH low dose
Other: Non-treatment control group
  Arms: PEG-rhGH high dose; PEG-rhGH low dose

SUMMARY:
This study aims to explore the optimal dose of pegylated recombinant human growth hormone (PEG-rhGH) injection to treat children of Turner syndrome (TS), preliminarily evaluate its safety and efficacy and provide scientific and reliable evidence for the medication dosage in Phase 3 clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Bone age <12 years
* Karyotype: 45, X; 45, X / 46, XXqi; 45, X / 46, XXr; 45, X / 46, XX; 46, XXqi; 46, XXpi; 45, X / 47, XXX; 46, XXp-; 45, X / 46, XXp-; 46, XXq-; 45X / 46, XXq-; 45, X / 46, XX / 47, XXX, etc. (count 50 or more cells);
* Facial appearance and abnormalities: Patients with at least one of the following signs, which include but are not limited to facial pigmented nevus, short neck, webbed neck, low posterior hairline, low-set ears, micrognathia, high-voulted arch, shield-like chest, cubitus valgus, genu valgum, short 4th and 5th metacarpals, nail dysplasia, scoliosis, ptosis and strabismus, cardiovascular abnormalities (such as aortic stenosis, bicuspid aortic valve and hypertension), reproductive abnormalities (such as primary gonadal dysfunction), renal abnormalities, thyroid hypofunction, middle ear lesion, etc.
* Short stature: height below -2.5SD of the mean height of the same age and gender.
* Pre-pubertal (Tanner Stage I ) patients
* No history of growth hormone treatment
* The subject and his/her guardian sign the informed consent (if the subject is incapable to sign the informed consent, his/her legal guardian shall sign the name of the subject instead)

Exclusion Criteria:

* Subjects with abnormal liver and kidney functions (ALT > upper limit of normal value; Cr > upper limit of normal value)
* Subjects positive for anti-HBc, HbsAg or HbeAg in Hepatitis B virus tests;
* Subjects with highly allergic constitution or allergy to proteins or investigational product or its excipient
* Subjects with systemic chronic disease and immune deficiency
* Patients diagnosed with tumor
* For patients whose tumor markers exceeding normal range in combination with other information, considering as potential high risks of tumor, they may be excluded from the treatment.
* Patients with mental disease
* Subjects with impaired glucose regulation (IGR) (including impaired fasting glucose (IFG) and/or impaired glucose tolerance (IGT) ) or diabetes
* Subjects who took part in other clinical trials within 3 months
* Subjects who received medicines which may interfere GH secretion or GH function, or other hormones within 3 months (such as sex steroids, glucocorticoids, etc.)
* Other conditions which are unsuitable for this study in the opinion of the investigator.

Ages: 2 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Change of height standard deviation score before and after treatment (ΔHT SDS) | 52 weeks
  The change of height standard deviation score of chronological age before and after treatment

SECONDARY OUTCOMES:
Height Velocity | 52 weeks
  Annual growth rate at the end of treatment
ΔBA/ΔCA | 52 weeks
  Bone maturation (changes of bone age/ chang of chronological age)
IGF-1(Insulin-like growth factor 1) SDS | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chunxiu Gong, PhD, Principal Investigator — Beijing Children's Hospital
Locations (9):
- China (9):
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Jiangxi Provincial Children's Hospital, Nanchang, Jiangxi
  - First Hospital of Jilin University, Changchun, Jilin
  - The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Beijing Children's Hospital,Capital Medical University, Beijing
  - Children's Hospital of Fudan University, Shanghai
  - Shanghai Children's Hospital, Shanghai
  - Xinhua Hospital of Shanghai Jiao Tong University School of Medicine, Shanghai